CLINICAL TRIAL: NCT03632824
Title: Tranexamic Acid for Antepartum Bleeding of Unknown Origin in the Second and Third Trimester: Nonrandomized Controlled Trials
Brief Title: Tranexamic Acid in Pregnancies With Vaginal Bleeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hawler Medical University (Other)
Responsible Party: Principal Investigator, Ariana Jawad, Assistant Professor, Hawler Medical University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HawlerMU 27.7
Record Dates: First submitted 2018-07-27; First posted 2018-08-15 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Vaginal Bleeding During Pregnancy
Keywords: Antepartum bleeding; Perinatal morbidity; Perinatal mortality; Preterm labor
MeSH Terms: conditions — Perinatal Death; Obstetric Labor, Premature | interventions — Tranexamic Acid

STUDY DESIGN:
Intervention Model Description: Tranexamic acid was prescribed for pregnant women with vaginal bleeding of unknown etiology in second and third trimester (13-34 weeks) gestation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- interventional arm (Experimental): Tranexamic acid applied intravenously for 2 days followed by oral tranexamic acid
  Interventions: Drug: Tranexamic Acid
- comparative group (Placebo Comparator): expectant management, including admission to hospital, ultrasound examination at least twice a week, regular blood coagulation tests, fetal wellbeing , frequent ultrasound performing for placenta location ,betamethasone administration for whom delivery was suspected
  Interventions: Drug: Tranexamic Acid

INTERVENTIONS:
Drug: Tranexamic Acid — One gram( 2 ampules ) of tranexamic acid was received by the participant intravenously twice daily for 48 hours followed by 500 mg tranexamic acid tablet three times daily for 5 days .
  follow up of the patient was done by recurrence of the bleeding latter on during pregnancy . the course of treatment was repeated again .
  Other Names: Trenaxa , Manufacturer Macleods Pharmaceuticals; TRANSAMIN , NIKOLAKOPOULOS A.E. GALATSIOU AVENUE, Athens

SUMMARY:
Tranexamic acid has been proposed and used for prevention and management of antepartum and postpartum hemorrhage.

DETAILED DESCRIPTION:
Bleeding during pregnancy is associated with a three- to fourfold increase in perinatal mortality. Hemorrhage in pregnancy is characterized by activation of the fibrinolytic system. Tranexamic acid is a potent pharmaceutical agent that suppresses fibrinolysis, and thus can be used for managing hemorrhage in pregnancy. The FDA's pregnancy category for tranexamic acid is category B. Tranexamic acid has been used to decrease blood loss and treatment of intra partum blood loss in cesarean section also it has been used for prevention and management of postpartum hemorrhage after vaginal bleeding, regardless of whether the bleeding is due to genital tract trauma or other causes.

ELIGIBILITY:
Inclusion Criteria:

* pregnant woman having vaginal bleeding
* Second and third trimester of unknown etiology
* No placenta previa, abruptio placentae, local cervical or vaginal causes for bleeding
* Primigraivid, multiparous and grand multiparous woman
* Accept to participate in the trial

Exclusion Criteria:

* Hypersensitivity to tranexamic acid
* Women with acquired defective color vision
* History of venous thromboembolism
* Refused to participate

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 139 (Estimated)
Dates: Start 2016-02-01 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2020-01-18 (Actual)

PRIMARY OUTCOMES:
Cessation of vaginal bleeding as self-reported by women | 7 days
  Following up the pregnant woman clinically to approve cessation of vaginal bleeding after Tranexamic acid use using yes/No format
Gestational age | up to 7 days postpartum
  Newborn delivered before, at or after 20 weeks gestation in weeks
Rate of perinatal deaths | 7 dya after delivery
  total number of newborn delivered showing no signs of life (movement, appearance, cardiac pulsation) plus deaths of newborn in first week of life
Neonatal Apgar(Appearance, Pulse, Grimace, Activity, and Respiration) score Apgar scores includes 10 sores , 2 for each . The Apgar score was classified as severely depressed <0-3>, moderately depressed<4-6> and excellent condition<7-10> | Up to fifth minutes of life
  Apgar scores includes 10 sores , 2 for each . The Apgar score was classified as severely depressed 0-3, moderately depressed 4-6 and excellent condition 7-10

CONTACTS AND LOCATIONS:
Overall Officials: Ariana K. Jawad, Principal Investigator — Hawler Medical University, college of Medicine, department of Obstetrics and Gynecology
Locations (1):
- Hawler Medical University, Erbil, Kurdistan Region, Iraq